CLINICAL TRIAL: NCT00543062
Title: Thorough QT/QTc Study of Staccato® Prochlorperazine for Inhalation in Healthy Volunteers
Brief Title: Staccato Prochlorperazine Thorough QT/QTc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-001-102; 20 July 2007
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2008-11

CONDITIONS: Cardiotoxicity
Keywords: Inhaled prochlorperazine, Thorough Qt/QTc,
MeSH Terms: conditions — Cardiotoxicity | interventions — Loxapine; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Female and male subjects in approximately equal numbers were randomly assigned (1:1:1:1) to receive the 4 treatment sequences
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This was a double-blind, double dummy, placebo controlled, randomized 4-period crossover study to assess the effects of single doses of 5 and 10 mg of Staccato Prochlorperazine on QT intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence ABCD (Other): Treatment Sequence ABCD where Treatment: A = Inhaled prochlorperazine (10 mg) + oral placebo, B = Inhaled prochlorperazine (5 mg) + oral placebo, C = Inhaled placebo + oral placebo, D = Inhaled placebo + oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled placebo; Drug: Oral placebo; Drug: Inhaled prochlorperazine 5 mg; Drug: Inhaled prochlorperazine 10 mg; Drug: Oral moxifloxacin
- Treatment Sequence BDAC (Other): Treatment Sequence BDAC where Treatment: A = Inhaled prochlorperazine (10 mg) + oral placebo, B = Inhaled prochlorperazine (5 mg) + oral placebo, C = Inhaled placebo + oral placebo, D = Inhaled placebo + oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled placebo; Drug: Oral placebo; Drug: Inhaled prochlorperazine 5 mg; Drug: Inhaled prochlorperazine 10 mg; Drug: Oral moxifloxacin
- Treatment Sequence CABD (Other): Treatment Sequence CABD where Treatment: A = Inhaled prochlorperazine (10 mg) + oral placebo, B = Inhaled prochlorperazine (5 mg) + oral placebo, C = Inhaled placebo + oral placebo, D = Inhaled placebo + oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled placebo; Drug: Oral placebo; Drug: Inhaled prochlorperazine 5 mg; Drug: Inhaled prochlorperazine 10 mg; Drug: Oral moxifloxacin
- Treatment Sequence DCBA (Other): Treatment Sequence DCBA where Treatment: A = Inhaled prochlorperazine (10 mg) + oral placebo, B = Inhaled prochlorperazine (5 mg) + oral placebo, C = Inhaled placebo + oral placebo, D = Inhaled placebo + oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled placebo; Drug: Oral placebo; Drug: Inhaled prochlorperazine 5 mg; Drug: Inhaled prochlorperazine 10 mg; Drug: Oral moxifloxacin

INTERVENTIONS:
Drug: Inhaled placebo — Inhaled Staccato placebo (0 mg)
Drug: Oral placebo — Oral placebo (identical to 400 mg moxifloxacin)
Drug: Inhaled prochlorperazine 5 mg — Staccato prochlorperazine 5 mg, single dose
  Other Names: ADASUVE
Drug: Inhaled prochlorperazine 10 mg — Inhaled prochlorperazine 10 mg, single dose
  Other Names: ADASUVE
Drug: Oral moxifloxacin — Oral moxifloxacin 400 mg, si/ngle dose

SUMMARY:
To assess the safety of Staccato Prochlorperazine on cardiac repolarization (QTc interval duration) at 2 dose levels compared to placebo in healthy volunteers.

DETAILED DESCRIPTION:
The planned study is a single dose, double-blind, double-dummy, active and placebo controlled, randomized, 4-period cross-over study investigating investigating 2 doses levels of Staccato Prochlorperazine, a positive control with known QT/QTc prolongation (oral moxifloxacin), and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 to 65 years, inclusive.
2. Body mass index (BMI) ≥21 and ≤30.
3. Subjects who are willing and able to comply with the study schedule and requirements, and stay at the CRU for a 3-day period and 3 consecutive 2-day periods.
4. Subjects who speak, read, and understand English and are willing and able to provide written informed consent on an IRB approved form prior to the initiation of any study procedures.
5. Subjects who are in good general health prior to study participation as determined by a detailed medical history, physical examination, 12-lead ECG, blood chemistry profile, hematology, urinalysis, and in the opinion of the Principal Investigator.
6. Female participants (if of child-bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) who agree to use a medically acceptable and effective birth control method throughout the study and for one week following the end of the study.

Exclusion Criteria:

1. Subjects who regularly consume large amounts of xanthine-containing substances must be excluded.
2. Subjects who have taken prescription or nonprescription medication within 5 days of Treatment Period 1 must be excluded.
3. Subjects who have had an acute illness within the last 5 days of Treatment Period 1 must be excluded.
4. Subjects who have smoked tobacco within the last year must be excluded.
5. Subjects who have a history of HIV positivity must be excluded.
6. Subjects who have a history of allergy or intolerance to prochlorperazine or phenothiazines must be excluded.
7. Subjects who have a history of contraindication to anticholinergics must be excluded.
8. Subjects who have a history of pheochromocytoma, seizure disorder, Parkinson's disease, or Restless Leg Syndrome must be excluded.
9. Subjects who have an ECG abnormality must be excluded.
10. Subjects who have a history within the past 2 years of drug or alcohol dependence or abuse as defined by DSM-4 must be excluded.
11. Subjects who have a history of syncope, unstable angina, myocardial infarction (within 6 months), congestive heart failure, transient ischemic attack, or pheochromocytoma must be excluded.
12. Subjects who have a history of asthma or chronic obstructive lung disease must be excluded.
13. Subjects who have hypotension (systolic ≤90 mmHg, diastolic ≤50 mmHg), or hypertension (systolic ≥140 mmHg, diastolic blood pressure ≥90 mmHg) must be excluded.
14. Subjects who test positive for alcohol or have a positive urine drug screen must be excluded.
15. Female subjects who have a positive pregnancy test at screening or during randomization visit, or are breastfeeding must be excluded.
16. Subjects who have received an investigational drug within 30 days prior to the Screening Visit must be excluded.
17. Subjects who are considered by the investigator, for any reason, to be an unsuitable candidate for receiving prochlorperazine, or unable to use the inhalation device, must be excluded.
18. Subjects who have any other disease(s), by history, physical examination, or laboratory abnormalities (ALT or AST > 2-fold the upper limit of normal, bilirubin > 1.5 mg/dL, or creatinine > 1.8 mg/dL) or that in the investigator's opinion present undue risk to the subject or may confound the interpretation of study results must be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall R Stoltz, MD, Principal Investigator — Covance GFI Research, Evansville, IN 47714
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects reported to the CRU for baseline assessments (Day 1). The subjects were confined to the Clinical Research Unit under continuous medical or paramedical observation until at least 24 hours after each dose of Staccato Prochlorperazine or placebo.
Groups:
- Treatment Sequence ABCD; Treatment Sequence BDAC; Treatment Sequence CABD; Treatment Sequence DCBA: All subjects were to receive all 4 treatments in this 4 treatment crossover
Period: Overall Study
Arm/Group | Treatment Sequence ABCD | Treatment Sequence BDAC | Treatment Sequence CABD | Treatment Sequence DCBA
Started | 12 | 12 | 12 | 12
Completed | 10 | 11 | 9 | 11
Not Completed | 2 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Safety Population: All subjects were to receive all 4 treatments in this 4 treatment crossover
Arm/Group | Safety Population
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Maximum Effect of Inhaled Prochlorperazine on Cardiac Repolarization (QTc Interval Duration) at the Maximum Clinical Dose Compared to Placebo
Description: Time-matched differences in QTcI values between the maximum of the mean difference from baseline of the QTcI interval after time-matched placebo subtraction for treatment at 11 post-inhalation times.
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 22 hr
Population: QT population -- LSM and CI statistics were based on the individual (within subject) corrected differences between prochlorperazine and placebo exposures per ICH Guideline E14 for a thorough QT/QTc study.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Placebo+Inhaled Prochlorperazine 5 mg Crossover Subjects: All subjects who completed both treatments B and C: Treatment: B = Inhaled prochlorperazine (5 mg) + oral placebo, C = Inhaled placebo + oral placebo
  The analyses are based on a within (paired) comparison of the time matched drug - placebo QTc values.
- Placebo+Inhaled Prochlorperazine 10 mg Crossover Subjects: All subjects who completed both treatments A and C: Treatment: A = Inhaled prochlorperazine (10 mg) + oral placebo, C = Inhaled placebo + oral placebo.
  The analyses are based on a within (paired) comparison of the time matched drug - placebo QTc values.
Arm/Group | Placebo+Inhaled Prochlorperazine 5 mg Crossover Subjects | Placebo+Inhaled Prochlorperazine 10 mg Crossover Subjects
Number analyzed (Participants) | 42 | 42
milliseconds | 5.493 [2.635 to 8.351] | 5.229 [2.405 to 8.052]

2. Secondary Outcome: QTcI Versus Prochlorperazine Concentration
Description: QTcI @ median prochlorperazine concentration (3.75 mcg/mL) based on linear and nonlinear regression of QTcI versus time matched serum prochlorperazine concentrations
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 22 hr
Population: 846 paired QTcI and prochlorperazine concentration pairs from 42 subjects receiving prochlorperazine (5 or 10 mg)
  Each measure was based on the individual (within subject) corrected differences between prochlorperazine and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Inhaled Prochlorperazine: Serum concentrations following Staccato prochlorperazine 5 and 10 mg, single dose
Arm/Group | Inhaled Prochlorperazine
Number analyzed (Participants) | 42
milliseconds | 2.83 [1.11 to 4.56]

3. Secondary Outcome: Numbers and % of Subjects With QTcI > 450 ms
Description: Numbers and Percents of Subjects with QTcI exceeding 450 ms
Time Frame: 24 hours
Population: QT Population (placebo and prochlorperazine only)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Inhaled placebo Oral placebo
  Inhaled placebo: Inhaled Staccato placebo (0 mg)
  Oral placebo: Oral placebo (identical to 400 mg moxifloxacin)
- Inhaled Prochlorperazine 5 mg: Staccato prochlorperazine 5 mg, single dose Oral placebo
  Oral placebo: Oral placebo (identical to 400 mg moxifloxacin)
  Inhaled prochlorperazine 5 mg: Staccato prochlorperazine 5 mg, single dose
- Inhaled Prochlorperazine 10 mg: Staccato prochlorperazine 10 mg, single dose Oral placebo
  Oral placebo: Oral placebo (identical to 400 mg moxifloxacin)
  Inhaled prochlorperazine 10 mg: Inhaled prochlorperazine 10 mg, single dose
Arm/Group | Placebo | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg
Number analyzed (Participants) | 44 | 44 | 46
Participants | 3 | 4 | 6

4. Secondary Outcome: Numbers and % of Subjects With QTcI > 480 ms
Description: Numbers and Percents of Subjects with QTcI exceeding 480 ms at any of the outcome measure time points
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 22 hr
Population: QT population -- LSM and CI statistics were based on the individual (within subject) corrected differences between active and placebo exposures per ICH Guideline E14 for a thorough
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Inhaled placebo + Oral placebo
- Inhaled Prochlorperazine 5 mg: Staccato prochlorperazine 5 mg, single dose Oral placebo
Arm/Group | Placebo | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg
Number analyzed (Participants) | 45 | 45 | 46
Participants | 0 | 0 | 1

5. Secondary Outcome: Numbers and % of Subjects With QTcI Change > 30 ms
Description: Numbers and Percents of Subjects with QTcI increase from baseline exceeding 30 ms at any of the outcome measure time points
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 22 hr
Population: QT population -- LSM and CI statistics were based on the individual (within subject) corrected differences between active and placebo exposures per ICH Guideline E14 for a thorough QT/QTc study.
Measure: Count of Participants; unit: Participants
Groups:
- Inhaled Prochlorperazine 5 mg: Staccato prochlorperazine 5 mg, single dose + Oral placebo
- Inhaled Prochlorperazine 10 mg: Inhaled prochlorperazine 10 mg: Inhaled prochlorperazine 10 mg, single dose + Oral placebo
Arm/Group | Placebo | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg
Number analyzed (Participants) | 43 | 44 | 46
Participants | 0 | 1 | 0

6. Secondary Outcome: Numbers and % of Subjects With QTcI Change > 60 ms
Description: Numbers and Percents of Subjects with QTcI increase from baseline exceeding 60 ms at any of the outcome measure time points
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 22 hr
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg
Number analyzed (Participants) | 43 | 44 | 46
Participants | 0 | 0 | 0

7. Other Pre Specified Outcome: Maximum Effect of Moxifloxacin on Cardiac Repolarization (QTc Interval Duration) Compared to Placebo (Study Assay Sensitivity)
Description: A thorough QT/QTc study may be considered to have demonstrated assay sensitivity if 1 or more of the lower 95% CI values exceeds 5 msec
Time Frame: 1, 1.5, 2, 2.5, 3, 5 hours
Population: QT population -- LSM and CI statistics were based on the individual (within subject) corrected differences between moxifloxacin and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliseconds
Groups:
- Placebo+Oral Moxifloxacin 400 mg Crossover Subjects: All subjects who completed both treatments C and D: Treatment: C = Inhaled placebo + oral placebo, D = Inhaled placebo + oral moxifloxacin 400 mg
  The analyses are based on a within (paired) comparison of the time matched drug - placebo QTc values.
Arm/Group | Placebo+Oral Moxifloxacin 400 mg Crossover Subjects
Number analyzed (Participants) | 42
milliseconds | 9.595 [6.062 to 13.128]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed predose and at 14 pre-specified time points as well as whenever spontaneously reported by the subjects or study staff
Groups:
- Oral Moxifloxacin 400 mg: Oral moxifloxacin 400 mg Inhaled placebo
  Inhaled placebo: Inhaled Staccato placebo (0 mg)
  Oral moxifloxacin: Oral moxifloxacin 400 mg, si/ngle dose
Arm/Group | Placebo | Inhaled Prochlorperazine 5 mg | Inhaled Prochlorperazine 10 mg | Oral Moxifloxacin 400 mg
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44 | 0/46 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44 | 0/46 | 0/43
Other Adverse Events (participants affected / at risk) | 4/45 | 24/44 | 29/46 | 4/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | Inhaled Prochlorperazine 5 mg (N=44) | Inhaled Prochlorperazine 10 mg (N=46) | Oral Moxifloxacin 400 mg (N=43)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4) | 6 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 13 (13) | 12 (12) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 9 (9) | 1 (1)

LIMITATIONS AND CAVEATS:
The use of healthy subjects precludes observation of drug-induced QTc prolongation in a population with additional factors predisposing to TdP. Subjects with respiratory disease were excluded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less